CLINICAL TRIAL: NCT00167739
Title: Short Course of Quinine Plus a Single Dose of Sulphadoxine-Pyrimethamine for Plasmodium Falciparum Malaria
Brief Title: Treatment of Malaria With Quinine Plus Sulfadoxine-Pyrimethamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Schweitzer Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04/2003/Q/SP
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Malaria
Keywords: Malaria; Quinine; Sulfadoxine-pyrimethamine; Gabon
MeSH Terms: conditions — Malaria | interventions — Quinine; fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: Quinine plus sulfadoxine-pyrimethamine

SUMMARY:
Quinine remains the treatment of choice of hospitalised malaria cases. The long treatment duration of 7 days, and adverse reactions often hamper its adequate use. Reducing the treatment duration by adding sulfadoxine-pyrimethamine may enhance compliance and reduce side effects.

The efficacy of a 3-day treatment of quinine plus sulfadoxine-pyrimethamine for the treatment of hospitalised, uncomplicated malaria cases was assessed.

DETAILED DESCRIPTION:
One main concern of clinicians in malaria endemic areas is to find a simple malaria treatment with short treatment duration. The concept of combination therapy, which may reduce treatment duration and delay the spread of drug resistance in addition to an increase in efficacy, has been therefore introduced.

In contrast to the outpatient treatment of malaria where emergence of resistance has lead to new drugs policies, the treatment of hospitalised malaria cases remains, in many endemic countries, intravenous quinine for 7 days. The efficacy of this regimen is well established throughout Africa. The effectiveness of the quinine treatment may be considerably lower because of discontinuation of treatment due to early discharge, the occurrence of side effects or because of the fact that patients feel better and stop the treatment. Therefore, sulfadoxine-pyrimethamine (SP) is often added at discharge. This regimen has been shown to be effective. But in Africa, where the practice seems widespread, it has been assessed in only two trials.

Since resistance of Plasmodium falciparum to SP is increasing rapidly in Africa and there is evidence that SP monotherapy induce gametocytaemia, we hypothesize that the combination quinine/SP increases SP efficacy and prevents induction of gametocytaemia. In addition, since the use of the full course of quinine therapy may be hampered by many factors (hospital cost, hospitalisation duration, availability of beds, compliance and side effects), the addition of the long acting SP to complete a short course of quinine treatment may prevent recrudescence or reinfection and may increase effectiveness of malaria treatment and reduce postdischarge morbidity.

The efficacy and safety of the short course of intravenous quinine (3-day treatment) plus a single dose of oral SP for the treatment of falciparum malaria was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated falciparum malaria
* Asexual parasitaemia between 20,000 and 200,000/µL
* No mixed plasmodial infection
* Fever with temperature above 38 °C or history of fever during the preceding 24 hours
* No effective anti-malarial treatment for the present attack
* Informed consent

Exclusion Criteria:

* Haemoglobin < 7 g/dL
* Packed-cell volume < 20%
* White cell count > 16,000/µL
* Platelet count < 40,000/µL
* Schizontaemia > 50/µL
* Impaired consciousness
* Convulsions or history of convulsions
* Concomitant diseases masking assessment of response

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2003-04; Study Completion 2004-02

PRIMARY OUTCOMES:
Proportion of cured patients by day 28

SECONDARY OUTCOMES:
Proportion of gametocytes carriers during the hospitalisation period and on days 7, 14, 21, and 28
Parasite clearance time
Fever clearance time
Assessment of adverse events during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Michel A. Missinou, PhD, Principal Investigator — Albert Schweitzer Hospital
Locations (1):
- Medical Research Unit, Lambaréné, Lambaréné, Moyen-Ogooué Province, Gabon

REFERENCES:
- [Background] Kremsner PG, Winkler S, Brandts C, Neifer S, Bienzle U, Graninger W. Clindamycin in combination with chloroquine or quinine is an effective therapy for uncomplicated Plasmodium falciparum malaria in children from Gabon. J Infect Dis. 1994 Feb;169(2):467-70. doi: 10.1093/infdis/169.2.467. PMID 8106787
- [Background] Alloueche A, Bailey W, Barton S, Bwika J, Chimpeni P, Falade CO, Fehintola FA, Horton J, Jaffar S, Kanyok T, Kremsner PG, Kublin JG, Lang T, Missinou MA, Mkandala C, Oduola AM, Premji Z, Robertson L, Sowunmi A, Ward SA, Winstanley PA. Comparison of chlorproguanil-dapsone with sulfadoxine-pyrimethamine for the treatment of uncomplicated falciparum malaria in young African children: double-blind randomised controlled trial. Lancet. 2004 Jun 5;363(9424):1843-8. doi: 10.1016/S0140-6736(04)16350-2. PMID 15183620
- [Background] Bousema JT, Gouagna LC, Meutstege AM, Okech BE, Akim NI, Githure JI, Beier JC, Sauerwein RW. Treatment failure of pyrimethamine-sulphadoxine and induction of Plasmodium falciparum gametocytaemia in children in western Kenya. Trop Med Int Health. 2003 May;8(5):427-30. doi: 10.1046/j.1365-3156.2003.01047.x. PMID 12753638
- [Background] Kremsner PG, Krishna S. Antimalarial combinations. Lancet. 2004 Jul 17-23;364(9430):285-94. doi: 10.1016/S0140-6736(04)16680-4. PMID 15262108
- [Background] Athan E, Durrheim DN, Barnes K, Mngomezulu NM, Mabuza A, Govere J. Effectiveness of short-course quinine and single-dose sulfadoxine-pyrimethamine in the treatment of Plasmodium falciparum malaria in Mpumalanga Province, South Africa. S Afr Med J. 2001 Jul;91(7):592-4. PMID 11544977
- [Background] Rahman MR, Paul DC, Rashid M, Ghosh A, Bangali AM, Jalil MA, Faiz MA. A randomized controlled trial on the efficacy of alternative treatment regimens for uncomplicated falciparum malaria in a multidrug-resistant falciparum area of Bangladesh--narrowing the options for the National Malaria Control Programme? Trans R Soc Trop Med Hyg. 2001 Nov-Dec;95(6):661-7. doi: 10.1016/s0035-9203(01)90108-7. PMID 11816441
- [Background] Ogutu BR, Nzila AM, Ochong E, Mithwani S, Wamola B, Olola CH, Lowe B, Kokwaro GO, Marsh K, Newton CR. The role of sequential administration of sulphadoxine/pyrimethamine following quinine in the treatment of severe falciparum malaria in children. Trop Med Int Health. 2005 May;10(5):484-8. doi: 10.1111/j.1365-3156.2005.01415.x. PMID 15860096
- [Background] Deloron P, Mayombo J, Le Cardinal A, Mezui-Me-Ndong J, Bruzi-Baert C, Lekoulou F, Elissa N. Sulfadoxine-pyrimethamine for the treatment of Plasmodium falciparum malaria in Gabonese children. Trans R Soc Trop Med Hyg. 2000 Mar-Apr;94(2):188-90. doi: 10.1016/s0035-9203(00)90272-4. PMID 10897366
- [Background] Hall AP, Doberstyn EB, Mettaprakong V, Sonkom P. Falciparum malaria cured by quinine followed by sulfadoxine-pyrimethamine. Br Med J. 1975 Apr 5;2(5961):15-7. doi: 10.1136/bmj.2.5961.15. PMID 1093610
- [Background] Hall AP, Doberstyn EB, Karnchanachetanee C, Samransamruajkit S, Laixuthai B, Pearlman EJ, Lampe RM, Miller CF, Phintuyothin P. Sequential treatment with quinine and mefloquine or quinine and pyrimethamine-sulfadoxine for falciparum malaria. Br Med J. 1977 Jun 25;1(6077):1626-8. doi: 10.1136/bmj.1.6077.1626. PMID 326337
- [Background] de Souza JM, Sheth UK, de Oliveira RM, Roulet H, de Souza SD. An open, randomized, phase III clinical trial of mefloquine and of quinine plus sulfadoxine-pyrimethamine in the treatment of symptomatic falciparum malaria in Brazil. Bull World Health Organ. 1985;63(3):603-9. PMID 3899397
- See also: General information on malaria at the website of the Malaria Foundation International — http://www.malaria.org
- See also: Homepage of the Medical Research unit, Lambarene — http://www.lambarene.org